CLINICAL TRIAL: NCT05222256
Title: Levosimendan Versus Adrenaline in Patients With Low Left Ventricular Function Undergoing Elective On-Pump Coronary Artery Bypass Graft Surgery. A Randomized Controlled Study
Brief Title: Comparison Between Levosimendan and Adrenaline in CABG Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelhafeez Ahmed, Assisstant lecturer of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tee in open heart surgery
Record Dates: First submitted 2021-12-06; First posted 2022-02-03 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Open Heart Surgery
MeSH Terms: interventions — Simendan; Epinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (L) levosimendan group (Experimental): Patients in this group will receive levosimendan (0.1 μg/kg/min) during re-warming of the patients.
  Interventions: Drug: Levosimendan
- Group (A) Adrenaline group (Active Comparator): Patients in this group will receive Adrenaline (0.05 μg /kg/min) during re-warming of the patients.
  Interventions: Drug: Adrenaline

INTERVENTIONS:
Drug: Levosimendan — Patients in this group will receive levosimendan
  Arms: Group (L) levosimendan group
Drug: Adrenaline — Patients in this group will receive Adrenaline
  Arms: Group (A) Adrenaline group

SUMMARY:
The aim of this study is to compare between levosimendan and adrenaline in patients with pre-existing impaired systolic function (EF 30-40%), undergoing elective on-pump CABG, as regards hemodynamics and echocardiographic parameters.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery are at risk of post-cardiotomy myocardial dysfunction. This condition causes delayed recovery, organ failure, prolonged intensive care unit and hospital stays, and an increased risk of mortality. These patients often require inotropic support, which has been associated with an increased risk of cardiovascular complications. Treatment of myocardial dysfunction includes optimization of myocardial contractility through appropriate fluid and pharmacologic management and mechanical support . Extensive use of inotropes in this situation is needed, but the optimal pharmacologic management of myocardial dysfunction in cardiac surgery is a matter of ongoing debate .Available inotropes including adrenaline may increase myocardial oxygen consumption, heart rate and risk of arrhythmia. An increase in myocardial oxygen consumption by inotropes in a state of inadequate oxygen delivery may further deteriorate underlying cardiac dysfunction and even lead to increased mortality . There are questions regarding the ideal inotrope to use during the post cardiopulmonary bypass (CPB) period in patients undergoing on-pump CABG surgery. The occurrence of myocardial dysfunction after cardiac surgery is a potential indication for the use of levosimendan, a calcium sensitizer with a unique mechanism of action. By binding to cardiac troponin C, it enhances myofilament responsiveness to calcium, thereby increasing myocardial contraction without increasing myocardial oxygen consumption. In addition, levosimendan activates adenosine triphosphate-dependent potassium channels, which are important mediators of ischemic and anesthetic cardioprotection. Levosimendan might thus have a potential benefit for patients with myocardial oxygen imbalance requiring inotropic drug support . The hypothesis of the present study is that levosimendan without loading dose can improve myocardial function and provide better hemodynamics as well as echocardiographic parameters compared with adrenaline in patients with low ejection fraction undergoing op-pump CABG

ELIGIBILITY:
Inclusion Criteria:

* ischemic hear disease
* age 18 and 65 years
* low left ventricular function (ejection fraction 30 - 40%),
* elective coronary artery bypass grafting (CABG) surgery

Exclusion Criteria:

* Age over 65 years
* Patients with end organ failure (renal, liver)
* Associated significant valve lesions
* Uncontrolled diabetes mellitus
* Emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Systolic function (EF) will be measured in both groups Levosemindan and Adrenaline in patients with low ejection fraction (30-40%), undergoing elective on pump Coronary Artery Bypass Graft (CABG). | 24 hour
  transesophageal echo (TEE) will be continuously used to monitor LV systolic and diastolic function during surgery and recordings will be made simultaneously with hemodynamic measurements. LV Ejection Fraction In the transgastric mid-papillary view, the echo machine will be switched to M-mode and the following measurements will be taken: o LV end-diastolic diameter o LV end-systolic diameter The machine will then calculate the LV ejection fraction according to Teich's method

SECONDARY OUTCOMES:
LV Myocardial Performance (Tei) Index will be measured in both groups | 24 hour
  The left ventricle myocardial performance index will be calculated by placing pulsed Doppler sample volume between the anterior leaflet of the mitral valve and the left ventricle outflow tract (LVOT) in the deep transgastric view. Tei index = (a-b)/b, where (a) = distance between the mitral A wave and E wave, and (b) = distance between the start and end of the LVOT flow)
LV Stroke Volume and Cardiac Output will be measured in both groups | 24 hour
  The LVOT diameter will be measured in the mid-esophagus long-axis view. Assuming that the LVOT is circular in shape, the LVOT cross-sectional area will be calculated . The velocity time integral (VTI) of LVOT will be determined by pulsed Doppler imaging in the deep transgastric view by tracing the LVOT ejection curve. The stroke volume (SV) will then be calculated as:
  Stroke volume (cm3) = LVOT cross sectional area x LVOT VTI
  Cardiac output (CO) will then be calculated as CO = SV x heart rate, and cardiac index (CI) will be calculated as CI = CO/body surface area.
LV diastolic function will be measured in both groups | 24 hour
  In the mid-esophageal four-chamber view, E-wave velocity, A-wave velocity and E/A ratio will be determined by placing the sample volume of pulsed-wave Doppler at the tips of the mitral leaflets. Using tissue Doppler imaging, e'-wave velocity will be measured at both the lateral and septal mitral annulus, and the average of both measurements will be reported and used in subsequent calculations. The E/e' index will be calculated